CLINICAL TRIAL: NCT01547520
Title: Meperidine as the Single Sedative Agent During Esophagogastroduodenoscopy, a Double-blind, Randomized Controlled Study
Brief Title: Meperidine as the Single Sedative Agent During Esophagogastroduodenoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dalin Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: DalinTCGH-hsieh-02
Record Dates: First submitted 2012-02-28; First posted 2012-03-08 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Esophagogastroduodenoscopy
Keywords: meperidine; esophagogastroduodenoscopy; unsedated; minimal sedation
MeSH Terms: interventions — Meperidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- meperidine (Experimental): 25 mg of meperidine is injected intramuscularly before EGD
  Interventions: Drug: Meperidine
- placebo (Placebo Comparator): placebo was given intramuscularly before EGD
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Meperidine — intramuscular, 25 mg, 5 to 10 minutes before EGD
  Arms: meperidine
Drug: normal saline — 25 ml of normal saline, intramuscular, 5 to 10 minutes before EGD
  Arms: placebo

SUMMARY:
Upper endoscopy is uncomfortable for most patients. Meperidine has both sedative and analgesic effects, so its use may be helpful for patients receiving upper endoscopy.

DETAILED DESCRIPTION:
Unsedated esophagogastroduodenoscopy (EGD) is a useful tool for upper gastrointestinal tract examination and therapy, but it is uncomfortable for many patients. Meperidine has been widely used in colonoscopic examination for many years; however, its use in EGD has not been completely evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing diagnostic upper endoscopy in our endoscopic room were enrolled.

Exclusion Criteria:

* A therapeutic upper endoscopic procedure, sedated endoscopy, contraindication to Buscopan (hyoscine N-butylbromide)
* Allergy to meperidine
* American Society of Anesthesiology (ASA) risk Class 3 or higher
* Renal failure
* Decompensated cirrhosis
* Aged less than 20 years or more than 65 years
* Pregnancy
* Refusal to provide written informed consent.

Ages: 20 Years to 65 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2011-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
discomfort score during esophageal intubation | 9 months
  patient self-reported discomfort score during esophageal intubation, assessed with a 0 to 10 visual analog scale (VAS)

SECONDARY OUTCOMES:
patient and endoscopist satisfaction score | 9 months
  patient and endoscopist satisfaction with the procedure, score 0(not satisfied at all)-10 (very satisfied
patient tolerance of the procedure | 9 months
  patolerace of the EGD, evaluate by the endoscopist, score 0 (best tolerance)-10 (very poor tolerance, the procedure could not be completed)
endoscopist perception of patient tolerance , | 9 months
  endoscopist evaluation of patient tolerance during EGD, score 0 (best tolerance)- 10 (worst tolerance, the procedure can not be completed)

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Hsi Hsieh, Dr., Principal Investigator — Dalin Tzu Chi General Hospital
Locations (1):
- Dalin Tzu Chi General Hospital, Chiayi City, Taiwan, Taiwan

REFERENCES:
- [Background] Abraham NS, Fallone CA, Mayrand S, Huang J, Wieczorek P, Barkun AN. Sedation versus no sedation in the performance of diagnostic upper gastrointestinal endoscopy: a Canadian randomized controlled cost-outcome study. Am J Gastroenterol. 2004 Sep;99(9):1692-9. doi: 10.1111/j.1572-0241.2004.40157.x. PMID 15330904
- [Background] Ishido S, Kinoshita Y, Kitajima N, Itoh T, Nishiyama K, Tojo M, Yano T, Inatome T, Fukuzaki H, Chiba T. Fentanyl for sedation during upper gastrointestinal endoscopy. Gastrointest Endosc. 1992 Nov-Dec;38(6):689-92. doi: 10.1016/s0016-5107(92)70565-3. PMID 1473671
- [Background] Laluna L, Allen ML, Dimarino AJ Jr. The comparison of midazolam and topical lidocaine spray versus the combination of midazolam, meperidine, and topical lidocaine spray to sedate patients for upper endoscopy. Gastrointest Endosc. 2001 Mar;53(3):289-93. doi: 10.1016/s0016-5107(01)70400-2. PMID 11231385
- [Background] Diab FH, King PD, Barthel JS, Marshall JB. Efficacy and safety of combined meperidine and midazolam for EGD sedation compared with midazolam alone. Am J Gastroenterol. 1996 Jun;91(6):1120-5. PMID 8651156
- [Derived] Hsieh YH, Lin HJ, Hsieh JJ, Tseng KC, Tseng CW, Hung TH, Leung FW. Meperidine as the single sedative agent during esophagogastroduodenoscopy, a double-blind, randomized, controlled study. J Gastroenterol Hepatol. 2013 Jul;28(7):1167-73. doi: 10.1111/jgh.12183. PMID 23431993